CLINICAL TRIAL: NCT05307042
Title: Decline in Renal Concentration Ability in Lithium Treated Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL72701.091.20
Record Dates: First submitted 2022-03-23; First posted 2022-04-01 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Lithium Toxicities; Bipolar Disorder; Concentration Ability Impaired; Nephrogenic Diabetes Insipidus; Lithium - Induced Nephropathy
MeSH Terms: conditions — Bipolar Disorder; Diabetes Insipidus, Nephrogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 2012-cohort
  Interventions: Diagnostic Test: Deamino Arginine Vasopressin (dDAVP)

INTERVENTIONS:
Diagnostic Test: Deamino Arginine Vasopressin (dDAVP) — After voiding, 40 μg 1-desamino-8-D arginine vasopressin (dDAVP) will be administered intranasally. Throughout the day, urine volume and maximal renal concentrating ability will be determined by measuring osmolality in urine collected at 4 and 6 hours after administration of dDAVP. In addition, water intake, body weight, blood pressure and heart rate will be determined at baseline and 6 hours after administration of dDAVP.

SUMMARY:
Lithium therapy is cornerstone in therapy of bipolar disorders. A well known side-effect of lithium therapy is a urinary concentration defect which manifests in it's most severe form as nephrogenic diabetes insipidus. The development of urinary concentration defects and its progression to nephrogenic diabetes insipidus in the population of lithium treated patients is unknown and therefore this study aims to evaluate the decline of urinary concentration defects in a Dutch population of lithium treated patients. In this prospective cohort study, 51 participants treated with lithium at Canisius Wilhelmina Hospital, Nijmegen and included in the previous study in 2012 will be approached to undergo a follow-up dDAVP-test.

ELIGIBILITY:
Inclusion Criteria:

* included in the previous study
* men and women
* age ≥ 18 years

Exclusion Criteria:

* General contra-indications for participation in a trial:

  * inability to give informed consent
  * pregnancy
  * unstable psychiatric condition
* Alternative causes of (nephrogenic) diabetes insipidus:

  * hypokalemia (plasma potassium < 3.0 mmol/l)
  * severe hypercalcemia (albumin-corrected plasma calcium > 2.80 mmol/l)
  * hyperglycemia (plasma glucose > 10.0 mmol/l)
  * history of amyloidosis, Sjögren's syndrome or Sickle cell anemia
  * previous treatment with ifosfamide
  * established primary polydipsia or central diabetes insipidus
* Contra-indications for dDAVP administration:

  * inability to comply with water restriction
  * renal insufficiency (GFR < 45 ml/min/1.73 m2)
  * hyponatremia (plasma sodium < 130 mmol/l)
  * instable angina pectoris
  * decompensated cardial insufficiency
* Other:

  * concomitant treatment with desmopressin or democlocycline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The 51 patients treated with lithium who were included in the previous study in 2012/2013, in which they were subject to a dDAVP test.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Decline renal concentration ability | 10 years
  To explore the decline in renal concentration ability (RCA) in a Dutch population of lithium treated patient. The primary endpoint is the percentual change in maximal urine osmolality.

SECONDARY OUTCOMES:
Relation between changes in kidney function and renal concentration ability | 10 years
  To determine the correlation between changes in kidney function and renal concentration ability
Relation between history of lithium-use and renal concentration ability | 10 years
  To determine the relationship between renal concentration ability and clinical parameters (duration of lithium therapy, plasma lithium concentration, baseline plasma creatinine, sodium and potassium concentration and baseline urinary osmolality) of lithium treated patients.
Chronic kidney disease | 10 years
  To determine the number of patients with chronic kidney disease at follow-up.
Decline in kidney-function | 10 years
  To explore the decline in kidneyfunction (expressed as eGFR, estimated by the CKD-EPI equation).

CONTACTS AND LOCATIONS:
Overall Officials: T. Nijenhuis, Principal Investigator — Radboud University Medical Center
Locations (1):
- Canisius Wilhelmina Ziekenhuis, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided